CLINICAL TRIAL: NCT01701102
Title: Optimal Dose of Spinal Mepivacaine Combined With Fentanyl For Knee Arthroscopy
Brief Title: Study to Find Optimal Dose of Local Spinal Anesthetic (Mepivacaine) Combined With Narcotic (Fentanyl) For Knee Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital for Special Surgery, New York (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 11140
Record Dates: First submitted 2012-01-04; First posted 2012-10-04 (Estimated); Results first posted 2016-03-10 (Estimated); Last update posted 2016-04-05 (Estimated); Status verified 2016-03

CONDITIONS: Arthroscopic Knee Surgery
MeSH Terms: interventions — Mepivacaine; Fentanyl

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- Mepivacaine 37.5 mg (Active Comparator)
  Interventions: Procedure: Mepivacaine
- Mepivacaine 30 mg plus fentanyl 10 µg (Active Comparator)
  Interventions: Procedure: Mepivacaine (30 mg) plus fentanyl
- Mepivacaine 27 mg plus fentanyl 10 µg (Active Comparator)
  Interventions: Procedure: Mepivacaine (27 mg) plus fentanyl
- Mepivacaine 24 mg plus fentanyl 10 µg (Active Comparator)
  Interventions: Procedure: Mepivacaine (24 mg) plus fentanyl

INTERVENTIONS:
Procedure: Mepivacaine (24 mg) plus fentanyl — Mepivacaine (24 mg) and fentanyl (10 µg)
  Arms: Mepivacaine 24 mg plus fentanyl 10 µg
Procedure: Mepivacaine (27 mg) plus fentanyl — Mepivacaine (27 mg) and fentanyl (10 µg)
  Arms: Mepivacaine 27 mg plus fentanyl 10 µg
Procedure: Mepivacaine (30 mg) plus fentanyl — Mepivacaine (30 mg) and fentanyl (10 µg)
  Arms: Mepivacaine 30 mg plus fentanyl 10 µg
Procedure: Mepivacaine — Mepivacaine 37.5 mg
  Arms: Mepivacaine 37.5 mg

SUMMARY:
Prolonged motor block and delayed ability to walk are limitations of spinal anesthesia in ambulatory (same-day) surgery. This can be improved by lowering the dose of local anesthetic (a medication that, when injected around nerves, blocks nerve conduction, resulting in numbness and weakness) used in the spine, but too low a dose can result in an incomplete block (inadequate anesthesia) in some patients. There is evidence that adding a low dose of fentanyl, a narcotic, to mepivacaine enhances the anesthetic effect. The purpose of this study is to determine the lowest dose of mepivacaine, a local anesthetic, when combined with fentanyl, for which spinal anesthesia is adequate for ambulatory knee arthroscopy.

ELIGIBILITY:
Inclusion Criteria:

* Subjects aged 18-60
* Patients scheduled for "simple" knee arthroscopies, including meniscectomy, debridement, and plica.

Exclusion Criteria:

* Subjects aged <18 or >60
* Subjects greater than 190 cm in height
* Patients scheduled for ligament reconstruction or surgery involving bone
* Daily use of narcotics for greater than one week pre-op

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 56 (Actual)
Dates: Start 2011-12; Primary Completion 2012-07 (Actual); Study Completion 2013-12 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital for Special Surgery, New York, New York, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Mepivacaine 37.5 mg: Mepivacaine (37.5 mg)
- Mepivacaine 30 mg Plus Fentanyl 10 µg: Mepivacaine plus fentanyl: Mepivacaine (30 mg) and fentanyl (10 µg)
- Mepivacaine 27 mg Plus Fentanyl 10 µg: Mepivacaine plus fentanyl: Mepivacaine (27 mg) and fentanyl (10 µg)
- Mepivacaine 24 mg Plus Fentanyl 10 µg: Mepivacaine plus fentanyl: Mepivacaine (24 mg) and fentanyl (10 µg)
Period: Overall Study
Arm/Group | Mepivacaine 37.5 mg | Mepivacaine 30 mg Plus Fentanyl 10 µg | Mepivacaine 27 mg Plus Fentanyl 10 µg | Mepivacaine 24 mg Plus Fentanyl 10 µg
Started | 22 | 6 | 10 | 18
Completed | 22 | 6 | 10 | 18
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Mepivacaine 37.5 mg; Mepivacaine 30 mg Plus Fentanyl 10 µg; Mepivacaine 27 mg Plus Fentanyl 10 µg; Mepivacaine 24 mg Plus Fentanyl 10 µg: Mepivacaine plus fentanyl: Mepivacaine (24 - 37.5 mg) and fentanyl (10 µg)
- Total: Total of all reporting groups
Arm/Group | Mepivacaine 37.5 mg | Mepivacaine 30 mg Plus Fentanyl 10 µg | Mepivacaine 27 mg Plus Fentanyl 10 µg | Mepivacaine 24 mg Plus Fentanyl 10 µg | Total
Number analyzed (Participants) | 22 | 6 | 10 | 18 | 56
Age, Continuous [Mean (Full Range); unit: years] | 41 [19 to 55] | 50 [42 to 57] | 46 [27 to 60] | 45 [19 to 60] | 44 [19 to 60]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 3 | 2 | 5 | 22
  Male | 10 | 3 | 8 | 13 | 34
Body Mass Index [Mean (Standard Deviation); unit: kg/(m^2)] | 26.3 (3.8) | 26.0 (4.3) | 28.5 (5.6) | 28.7 (4.8) | 27.4 (4.6)

OUTCOME MEASURES:

1. Primary Outcome: Time From Spinal Administration to Block Regression to the S1 Dermatome in Post-Anesthesia Care Unit (PACU)
Description: The time frame of the study for each patient only covers the period between time of surgery and time of discharge from the hospital, which is on the same day as the day of surgery
Time Frame: Participants will be followed for the duration of their recovery after surgery in the post-anesthesia care unit (PACU), an expected average of 2-4 hours.
Measure: Median (Inter-Quartile Range); unit: minutes
Arm/Group | Mepivacaine 37.5 mg | Mepivacaine 30 mg Plus Fentanyl 10 µg | Mepivacaine 27 mg Plus Fentanyl 10 µg | Mepivacaine 24 mg Plus Fentanyl 10 µg
Number analyzed (Participants) | 22 | 6 | 10 | 18
minutes | 203 [165 to 231] | 195 [175 to 210] | 156 [135 to 180] | 159 [135 to 194]

ADVERSE EVENTS:
Arm/Group | Mepivacaine 37.5 mg | Mepivacaine 30 mg Plus Fentanyl 10 µg | Mepivacaine 27 mg Plus Fentanyl 10 µg | Mepivacaine 24 mg Plus Fentanyl 10 µg
Serious Adverse Events (participants affected / at risk) | 0/22 | 0/6 | 0/10 | 0/18
Other Adverse Events (participants affected / at risk) | 0/22 | 0/6 | 0/10 | 0/18

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes